CLINICAL TRIAL: NCT04856475
Title: An Open Label Phase II Study to Evaluate Neratinib for Treatment and Prevention of Subsequent CNS Event(s) in Patients With Brain Metastasis of Advanced HER2 Positive Breast Cancer
Brief Title: Evaluation of Neratinib for Treatment and Prevention of Subsequent CNS Event(s) in Patients With Brain Metastasis of Advanced HER2 Positive Breast Cancer
Acronym: NeraBrain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of collaboration with PUMA
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJB-NERABRAIN-ODN-007
Record Dates: First submitted 2021-03-30; First posted 2021-04-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — neratinib

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomised, phase II study to evaluate the efficacy of neratinib in combination with SOC systemic therapy on CNS metastasis both as for secondary prevention (cohort 1), primary treatment (cohort 2) and for the treatment of LM disease (cohort 3) in subjects with HER2 positive metastatic BC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HER2 metastatic breast cancer locally pretreated for previous CNS events and currently progressive (Experimental): Eligible subjects will receive neratinib in combination with capecitabine or with T-DM1 or with paclitaxel or with vinorelbine as per investigator's choice. Trastuzumab can be added as per investigator's choice to those regimens except for T-DM1.
  At screening and during the study treatment period (every 9 weeks), brain MRI and tumour assessment by thoracic and abdomino-pelvic CT scan should be performed. Additionally, at screening and at each cycle during the study treatment period, subjects must fill quality of life questionnaires: EORTC core questionnaire (QLQ-C30) and brain module (QLQ-BN20).
  Interventions: Drug: Neratinib
- HER2 positive metastatic breast cancer patients with newly diagnosed brain metastases (Experimental): Eligible subjects will receive neratinib in combination with capecitabine or with T-DM1 or with paclitaxel or with vinorelbine as per investigator's choice. Trastuzumab can be added as per investigator's choice to those regimens except for T-DM1.
  At screening and during the study treatment period (every 9 weeks), brain MRI and tumour assessment by thoracic and abdomino-pelvic CT scan should be performed. Additionally, at screening and at each cycle during the study treatment period, subjects must fill quality of life questionnaires: EORTC core questionnaire (QLQ-C30) and brain module (QLQ-BN20).
  Interventions: Drug: Neratinib
- HER2 positive metastatic breast cancer patients with leptomeningeal carcinomatosis (Experimental): Eligible subjects will receive neratinib in combination with capecitabine or with T-DM1 or with paclitaxel or with vinorelbine as per investigator's choice. Trastuzumab can be added as per investigator's choice to those regimens except for T-DM1.
  At screening and during the study treatment period (every 9 weeks), contrast-enhanced neuraxis brain and spine MRI and tumour assessment by thoracic and abdomino-pelvic CT scan should be performed. CSF cytological assessment should also be performed.
  Additionally, at screening and at each cycle during the study treatment period, subjects must fill quality of life questionnaires: EORTC core questionnaire (QLQ-C30) and brain module (QLQ-BN20).
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — As per investigator's choice, eligible subjects in all cohort will receive:
  * Neratinib, administered continuously at a dose of 240 mg orally once a day in combination with:
    * Capecitabine, administered continuously at a dose of 750 mg/m2, orally, twice a day (=daily dose of 1500 mg/m2) from D1 toD14 (21 days cycle) (preferred option) or
    * Vinorelbine, I.V. 25 mg/m2 on D1 and D8 (21 days cycle) or
    * Paclitaxel, I.V. 80 mg/m2 on D1, D8, and D15 (21 days cycle) Important note: The possibility to combine trastuzumab, loading dose 8 mg/kg IV followed by 6 mg/kg Q3W IV or SC 600 mg Q3W, to one of these above treatments is left at investigator's discretion OR
  * Neratinib, administered continuously at a dose of 160 mg, orally, once a day in combination with:
    * T-DM1, I.V. 3.6mg/m2 on D1 (21 days cycle) (preferred option)

SUMMARY:
This is an open-label, non-randomised, phase II study to evaluate the efficacy of neratinib in combination with SOC systemic therapy on CNS metastasis both as for secondary prevention (cohort 1), primary treatment (cohort 2) and for the treatment of LM disease (cohort 3) in subjects with HER2 positive metastatic BC.

Subjects with metastatic HER2 positive breast cancer will be eligible for the trial and will be enrolled in one of the following cohorts:

Cohort 1: Eligible subjects include HER2 positive metastatic breast cancer subjects treated with at least one line of systemic anti HER2 therapy and pre-treated with local approaches at least for the previous CNS event and currently progressive but locally treated CNS metastasis. Local therapy includes: stereotactic radiosurgery (SRS) or/and WBRT or/and surgery.

The study will measure the effect of the drug combination on the time to next CNS event(s).

Cohort 2: Eligible subjects include HER2 positive metastatic breast cancer subjects treated with at least one line of systemic anti HER2 therapy or progressing less than 12 months after end of adjuvant therapy with a first diagnosis of brain metastases.

The study will measure the objective CNS response in each subject.

Cohort 3: Eligible subjects include HER2 positive metastatic breast cancer subjects treated with at least one line of systemic anti HER2 therapy with confirmed LM defined as the presence of malignant cells in the cerebrospinal fluid (CSF) or combination of typical symptoms and MRI.

The study will measure the effect of the drug combination on the time to CNS progression including LM progression.

As per investigator's choice, eligible subjects in all cohort will receive neratinib in combination with capecitabine or with T-DM1 or with paclitaxel or with vinorelbine as per investigator's choice. Trastuzumab can be added as per investigator's choice to those regimens except for T-DM1.

At screening and during the study treatment period (every 9 weeks), brain MRI for cohort 1 and cohort 2 or contrast-enhanced neuraxis brain and spine MRI for cohort 3 and tumour assessment by thoracic and abdomino-pelvic CT scan for all cohorts should be performed. For cohort 3 only, CSF cytological assessment should also be performed.

Additionally, at screening and at each cycle during the study treatment period, subjects must fill quality of life questionnaires: EORTC core questionnaire (QLQ-C30) and brain module (QLQ-BN20).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status ≤ 2
3. Female
4. Diagnosis : histologically or cytologically confirmed HER2-positive tumour status according to the ASCO-CAP guidelines (defined as a 3+ score on immunohistochemistry (IHC) and/or positive by in situ hybridisation (ISH)) with brain metastases, estrogen receptor and progesteron receptor status Cohort 1: with CNS metastases pre-treated with local approaches for the previous CNS events and currently progressive but locally treated CNS metastasis Cohort 2: with a first diagnosis of CNS metastases, asymptomatic or paucisymptomatic not needing immediate local therapy Cohort 3: with confirmed LM defined as the presence of malignant cells in the CSF or combination of typical symptoms and MRI findings
5. Specific criteria for cohorts 1 and 2 only: Must have radiologically confirmed metastatic brain lesion by MRI measurable by RANO-BM criteria
6. Specific criteria for cohort 3 only: LM defined as the presence of malignant cells in the CSF or combination of typical symptoms and MRI findings for cohort 3
7. Subjects should have received at least 1 previous line for the metastatic disease including taxanes based chemotherapy in combination with trastuzumab and pertuzumab (if available) unless contraindicated. Prior tucatinib is not an exclusion criteria.
8. Corticosteroids may be used as long as subjects are on a stable or decreasing dose for at least 7 days prior to study enrolment
9. Serum pregnancy test (for subjects of childbearing potential) negative within 7 days prior to first neratinib administration
10. Women of childbearing potential must agree to use 1 highly effective or 2 effective methods of contraception (as defined at the protocol section 6.8.1) during the course of the study and at least 7 months after the last administration of study treatment.
11. Adequate bone marrow function as defined below:

    * Absolute neutrophil count ≥1500/µL or 1.5x109/L
    * Hemoglobin ≥ 9 g/dL
    * Platelets ≥100000/µL or 100x109/L
12. Adequate liver function as defined below:

    * Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome < 3 x ULN is allowed
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN (except in case of liver metastases AST/ALT ≤ 5 x ULN)
13. Adequate renal function as defined below:

    • Creatinine ≤ 1.5 x UNL or creatinine clearance >60 mL/min
14. Signed Informed Consent form (ICF) obtained prior to any study related procedure
15. LVEF > 55% Inclusion criterion applicable to FRANCE only 1)16) Affiliated to the French Social Security System

Exclusion Criteria:

1. CNS disease requiring immediate neurosurgical intervention (e.g. resection, shunt placement, etc.)
2. Any unresolved toxicity ≥ CTCAE grade 2 (except alopecia) from previous anti-cancer therapy
3. Is ineligible for or has already received all chemotherapy options among the physician's choice
4. Any evidence of severe or uncontrolled systemic disease such as clinically significant cardiovascular, pulmonary, hepatic, renal or metabolic disease
5. Specific criteria for cohort 2 only: Previous local treatment for CNS metastases
6. Specific criteria for cohort 2 only: Oligometastatic disease restricted to the CNS and for which a local treated is considered as the most appropriate treatment by the investigator.
7. Known DPD deficiency* tested by measuring the level of uracil in the blood, or by checking for the presence of certain mutations in the gene for DPD according to EMA recommendation in case investigator's choice is capecitabine
8. Received an investigational anti-cancer drug within four weeks or five half-lives (whichever is shorter) of study drug administration
9. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs
10. Known HIV, Hepatitis B or Hepatitis C infection
11. Pregnant and/or lactating women
12. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study
13. Contra-indication for contrast-enhanced MRI (either hypersensitivity to Gd chelate or absolute contra-indication for MRI such as non compatible cardiac stimulator) * Testing of subjects for DPD deficiency in case of capecitabine is proposed according to local practices Exclusion criterion applicable to FRANCE only Vulnerable persons according to the article L.1121-6 of the Public Health Code, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the Public Health Code

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
For cohort1: Efficacy of neratinib in combination with systemic treatment at investigator's choice in preventing the next CNS event in HER2 breast cancer with known and treated brain metastasis | From date of enrolment until the date of subsequent documented CNS event, assessed up to 6 months
  The efficacy will be assessed by calculating the ratio of the time to the subsequent CNS event (T2) according to RANO-BM criteria to the time between the current CNS event and previous CNS event (T1) both treated locally (T2/T1).
  The subsequent CNS event is defined as progression of known and treated brain lesions as well as the development of new brain lesions as assessed on magnetic resonance imaging (MRI) using the RANO-BM criteria.
  The time to a subsequent CNS event is defined as the time from treatment start of a CNS event to the occurrence of the following one for both T1 and T2
For cohort 2: Efficacy of neratinib in combination with systemic treatment at investigator's choice on previously untreated brain metastasis from HER2 metastatic breast cancer | From date of enrolment until the date of first documented CNS event, assessed up to 6 months
  The efficacy will be assessed by calculating the proportion of subjects with an objective CNS response, according to RANO-BM criteria in the absence of progressive extra-CNS disease (according to RECIST 1.1).
For cohort 3: Efficacy of neratinib in combination with systemic treatment at investigator's choice on LM disease from HER2 metastatic breast cancer | From date of enrolment until the date of first documented leptomeningeal progression or date of death from any cause, whichever came first, assessed up to 6 months
  The efficacy will be assessed by measuring CNS progression-free survival defined as the time between treatment start and date of first leptomeningeal progression (defined according to clinical-neurological or imaging criteria) in the absence of progressive extra-CNS disease (according to RECIST 1.1) or date of death (death from any cause) whatever occurs first.

SECONDARY OUTCOMES:
Efficacy of neratinib in combination with systemic treatment according to investigator's choice on brain metastasis | From date of enrolment until the date of next documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Occurrence of new brain metastases according to RECIST 1.1
For cohort 2 only: Evaluation of the time to the first CNS local treatment | From date of enrolment until the date of first documented CNS event, assessed up to 6 months
  Mesure of the time to the first CNS local treatment
Efficacy of neratinib in delaying the time to whole brain radiotherapy (WBRT) in HER2 breast cancer with known brain metastasis (for subject not previously submitted to WBRT) | From date of enrolment until the date of next documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Mesure of the time to whole brain radiotherapy (WBRT)
Safety of neratinib | Assessed up to 6 months
  Evaluation of the adverse events
Evaluation of the overall survival (OS) | up to 2 years
  Mesure of the number of overall survival
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Clinical Benefit (CB) according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Objective Response Rate (ORR) - including intracranial ORR according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Best Response (BR) according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of CNS Progression-Free survival according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Extra CNS Progression-Free survival. Assessment of extra-CNS lesions will use the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of overall Progression-Free Survival (PFS) according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Duration of Response (DoR) according to RANO-BM criteria and RECIST 1.1
Brain, systemic and bi-comportemental efficacy | Through study completion, up to 2 years
  Mesure of Duration of Clinical Benefit (DCB) according to RANO-BM criteria and RECIST 1.1
Assessment of the quality of life | Assessed up to 6 months
  Analysis of Quality of life questionnaire "EORTC QLQ-C30"
Assessment of the quality of life | Assessed up to 6 months
  Analysis of Quality of life questionnaire "Brain module QLQ-BN20"

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Kotecki, MD, Study Chair — Jules Bordet Institute

IPD SHARING:
Plan to Share IPD: Undecided